CLINICAL TRIAL: NCT05739682
Title: The Effect of Final Irrigation Using Antimicrobial-corticosteroid Mixture Versus Cryotherapy on Post-instrumentation Pain and Microbial Reduction in Patients Having Single Canal - Teeth With Necrotic Pulps: A Randomized Clinical Trial
Brief Title: Pain and Microbial Reduction of Antimicrobial Corticosteroid Mixture Versus Cryotherapy in Necrotic Teeth
Acronym: MIXCRYO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Fawzy Omar Mohammed Habib, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO 18-11-21
Record Dates: First submitted 2021-11-18; First posted 2023-02-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-02

CONDITIONS: Dental Pulp Necrosis
Keywords: Antibiotic; Antifungal; Corticosteroid; Cryotherapy
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Carticaine; Epinephrine; Root Canal Preparation; Root Canal Obturation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Both final irrigating solutions are colorless and will be delivered inside the root canal using a plastic syringe without the patient knowing the type of solution used.
  The microbial samples will be sent to the lab for microbial count assessment with a code without identification of the type of irrigating solution used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antimicrobial Corticosteroid mixture (Experimental): Each canal will receive 5 minutes of final irrigation with the antimicrobial-corticosteroid solution of a freshly prepared mixture of:
  1 ml of Levofloxacin (Tavanic, Sanofi Aventis, Egypt).
  1 ml of Fluconazole (Sunny fungal, Sunny pharmaceuticals, Egypt).
  1 ml of Dexamethasone sodium phosphate (Dexamethasone, Amriya, Egypt).
  Interventions: Procedure: Local anaesthetic injection of 4% articaine with 1:100000 epinephrine; Procedure: Tooth isolation; Procedure: Access cavity preparation; Procedure: Root canal shaping and cleaning; Procedure: Final irrigation with antimicrobial-corticosteroid mixture; Procedure: Temporary restoration and patient's instructions; Procedure: Root canal obturation
- Cryotherapy (Active Comparator): Each canal will receive final irrigation with 20ml of cold saline (2.5°c) for 5 minutes.
  Interventions: Procedure: Local anaesthetic injection of 4% articaine with 1:100000 epinephrine; Procedure: Tooth isolation; Procedure: Access cavity preparation; Procedure: Root canal shaping and cleaning; Procedure: Final irrigation with cold saline; Procedure: Temporary restoration and patient's instructions; Procedure: Root canal obturation

INTERVENTIONS:
Procedure: Local anaesthetic injection of 4% articaine with 1:100000 epinephrine — Buccal infiltration injection using a side loading aspirating syringe and a 30-gauge needle
Procedure: Tooth isolation — Rubber dam application to the affected tooth
Procedure: Access cavity preparation — Complete removal of caries, undermined tooth structure, and defective restoration. Access cavity preparation with complete removal of the pulp chamber roof using a sterile bur other than the ones used for caries removal.
Procedure: Root canal shaping and cleaning — Working length determination using an electronic apex locator and then canal instrumentation using Hyflex CM rotary files up to size 40.04 with irrigation using 2.5% NaOCl between files.
Procedure: Final irrigation with antimicrobial-corticosteroid mixture — 1 ml of levofloxacin will be withdrawn in a 3ml plastic syringe followed by 1 ml of fluconazole and 1 ml of dexamethasone sodium phosphate, the whole solution is then passively delivered into the canal using a 30-gauge side vented needle reaching 1 mm shorter than the working length. The solution will be left inside the canal for 5 minutes
  Arms: Antimicrobial Corticosteroid mixture
Procedure: Final irrigation with cold saline — Frozen sterile saline will be brought at room temperature and monitored using a digital liquid thermometer till the temperature reaches 2.5°c. 4ml are then withdrawn in a 5ml plastic syringe and delivered inside the canal in 1 minute. The process is then repeated 5 times so that the canal receives 20 ml of 2.5°c cold saline for 5 minutes.
  Arms: Cryotherapy
Procedure: Temporary restoration and patient's instructions — The canals are dried using paper points and the access cavity is sealed using a non-eugenol temporary filling.
Procedure: Root canal obturation — After the 1st visit by 3 days to 1 week, the patient is scheduled for a second appointment for root canal obturation.

SUMMARY:
The aim of this study is to compare the effect of antimicrobial-corticosteroid mixture and cryotherapy as final root canal irrigating solutions on post-instrumentation pain in single-canal teeth with necrotic pulps.

DETAILED DESCRIPTION:
The trial participants are patients with single-canal teeth with necrotic pulps undergoing root canal treatment on two visits. During the 1st visit, access cavity, root canal cleaning and shaping using rotary files and 2.5% NaOCl irrigation. After apical preparation, a final flush with either a levofloxacin-fluconazole-dexamethasone mixture or cold saline will be used then the tooth access cavity will be sealed with a temporary filling. After the first visit, the participants will be given a pain chart with a numerical rating scale to rate their pain levels from zero to 10 at 6, 12, 24, and 48 hours. Three microbial swabs will be collected for each participant: before instrumentation (S1), after instrumentation before final irrigation (S2), and after final irrigation (S3). After collecting data from all participants, statistical analysis will be conducted to compare the pain intensity and microbial load reduction percentages between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in good physical health; American Society of Anesthesiologists class I or II.
2. Patients whose age ranges between 18 and 50 years.
3. Male and female patients.
4. Patients having a single canal-tooth with necrotic pulp.
5. Patients who can understand the number rating scale (figure).
6. Patients who accept to participate in the trial and can sign the informed consent (figure).

Exclusion Criteria:

1. Pregnant females.
2. Patients with swelling.
3. Patients whose tooth is non-restorable.
4. Teeth with open apices.
5. Teeth with radiographic evidence of root resorption.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-02-09 (Actual)

PRIMARY OUTCOMES:
Postinstrumentation pain | At 6 hours after the 1st visit
  Pain as reported by the patient on a Numerical rating scale from 0 to 10 where 0 indicates no pain and 10 indicates the worst possible pain
Postinstrumentation pain | At 12 hours after the 1st visit
  Pain as reported by the patient on a Numerical rating scale from 0 to 10 where 0 indicates no pain and 10 indicates the worst possible pain
Postinstrumentation pain | At 24 hours after the 1st visit
  Pain as reported by the patient on a Numerical rating scale from 0 to 10 where 0 indicates no pain and 10 indicates the worst possible pain
Postinstrumentation pain | At 48 hours after the 1st visit
  Pain as reported by the patient on a Numerical rating scale from 0 to 10 where 0 indicates no pain and 10 indicates the worst possible pain

SECONDARY OUTCOMES:
Anti bacterial effect | At 24 hours after the 1st visit
  percentage of bacterial reduction after final irrigation as compared to after instrumentation.
  Cultures from collected paper points will be inoculated in sterile brain heart infusion (BHI) broth vials which will be dispersed with vortex for 30 seconds. The sterile BHI broth solution will then be serially diluted one-tenth dilution and plated onto the blood agar medium and incubated at 37°C aerobically for 24 hours. The resultant bacterial growth will be quantified by evaluating the number of colonies on the agar medium & the number of CFU/ml of each dilution will be calculated for each sample.
Antifungal effect | At 48 hours after the 1st visit
  Percentage of Candidal reduction after final irrigation as compared to after instrumentation.
  Cultures from collected paper points will be inoculated in sterile brain heart infusion (BHI) broth vials which will be dispersed with vortex for 30 seconds. The sterile BHI broth solution will be serially diluted one-tenth dilution and plated onto Sabouraud dextrose agar medium and incubated at 25°C aerobically for 48 hours. The resultant candida growth will be quantified by evaluating the number of colonies on the agar medium & the number of CFU/ml of each dilution will be calculated for each sample.

CONTACTS AND LOCATIONS:
Overall Officials: Maged M Negm, Professor in Endodontics, Study Chair — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Yes
We are planning to share individual patient's data regarding age, gender, preoperative pain score and outcome data
Supporting Information: Study Protocol, SAP
Time Frame: From 1/6/2024 - Forever
Access Criteria: Anyone with the link can view the supporting information
URL: https://drive.google.com/drive/folders/11vjiC0a6uQFZXT8EdRE7b0rfweak2GRk